CLINICAL TRIAL: NCT05667532
Title: The C-MERIT Screening Cohort: Contrast-enhanced Mammography for Breast Cancer Screening and Risk Assessment in Women With Dense Breasts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-0651; NCI-2022-10200 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-30; First posted 2022-12-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast Enhanced Mammography (Experimental)
  Interventions: Diagnostic Test: Contrast Enhanced Mammography

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Mammography — Screening Modality

SUMMARY:
To learn whether a new imaging technology, Contrast-Enhanced Mammography (CEM), compared to standard mammography, can better detect breast cancers in women with dense breasts

DETAILED DESCRIPTION:
Primary Objectives:

* To establish a cohort of 1,000 female MDACC patients with dense breasts who undergo screening contrast-enhanced mammography.
* To establish a comprehensive integrated database of imaging, clinical data, health measurements, and questionnaire data including data from the companion protocol PA17-0584.

Secondary Objectives:

* To perform within-subject comparison of the cancer detection rate between CEM and FFDM.
* To perform within-subject comparison of the sensitivity, specificity, and recall rates of CEM compared to low-energy (LE) images (FFDM equivalent) and compared to a combination of LE and DBT images among women with dense breasts.
* To evaluate the effect of the availability of prior imaging for comparison on the recall rates of CEM, FFDM and DBT.
* In patients who undergo screening breast ultrasound as a standard of care, to evaluate the performance of screening ultrasound for breast cancer detection and compare it with other imaging modalities of CEM, LE images, and DBT.

Exploratory Objectives:

* To combine imaging, blood biomarkers, health measurements and questionnaire data for assessment of breast cancer risk.
* To evaluate if the intensity of background parenchymal enhancement on CEM predicts breast cancer risk in women with dense breasts.
* To evaluate if patients consider CEM as a potentially acceptable imaging modality for routine breast cancer screening.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 30-75 years of age with dense breasts (ACR BI-RADS categories C and D) who undergo routine yearly mammography at participating MDACC sites
2. Willingness to co-enroll or currently enrolled in PA17-0584
3. Willingness to participate in the study and ability to provide informed consent

Exclusion Criteria:

1. Self-reported new breast symptoms since last mammogram including nipple discharge, palpable mass, skin dimpling, or focal pain.
2. Current or recent (within the prior 6 months) history of pregnancy or breast feeding
3. Personal history of breast cancer (DCIS or invasive breast cancer)
4. Treatment of any other type of cancer within the past 5 years excluding in-situ cervical and non-melanoma skin cancer
5. Breast biopsy within 6 months
6. Breast surgery within 12 months
7. Breast MRI, MBI, or CEM performed within 24 months
8. Known allergy to iodine-containing contrast agents
9. History of anaphylactic reaction to any substance that required hospitalization or IV placement in a patient with no known prior uneventful exposure to iodine-based IV contrast
10. Renal insufficiency (as defined by UTMDACC policy 3.30- attachment 1 (appendix D)

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify female MDACC patients with dense breasts who undergo contrast-enhanced mammography | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Olena Weaver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org